CLINICAL TRIAL: NCT02303028
Title: A Phase I and Enrichment Study of Low-dose Metronomic Topotecan and Pazopanib in Pediatric Patients With Recurrent or Refractory Solid Tumours
Brief Title: Phase I Dose Escalation Study of Topotecan and Pazopanib in Children With Recurrent/Refractory Solid Tumours
Acronym: TOPAZ
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: C17 Council (Other)
Responsible Party: Principal Investigator, Jim Whitlock, Chief, Division of Haematology/Oncology, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000046233; IND.217 (Other: NCIC CTG)
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Solid Tumors
Keywords: Pediatric; Solid Tumour
MeSH Terms: interventions — Topotecan; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topotecan and Pazopanib (Experimental): Low dose Topotecan will be given metronomically in combination with Pazopanib at the dose level assigned at study entry
  Interventions: Drug: Topotecan and Pazopanib

INTERVENTIONS:
Drug: Topotecan and Pazopanib — Low-dose metronomic Topotecan and Pazopanib will be escalated as per the dose escalation schema.
  Other Names: Hycamtin; Votrient

SUMMARY:
This is a phase I, dose escalation study where topotecan will be administered at lower doses given more frequently on a prolonged schedule (low dose metronomic; LDM), in combination with pazopanib administered in a specific dose range. The maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) will be evaluated for LDM topotecan in combination with pazopanib in children with recurrent or refractory solid tumours. Pharmacokinetic and pharmacodynamic studies will be conducted to further define the exposure to and activity of LDM topotecan in combination with pazopanib.

ELIGIBILITY:
INCLUSION:

1. Disease: Part 1-Relapsed or refractory solid tumours with histological verification of malignancy. Patients with CNS tumours are not eligible. Parts 2A and 2B - histological verification of one of the following solid tumours: Neuroblastoma or Rhabdomyosarcoma
2. Measurable or evaluable disease
3. No known curative therapy, or therapy proven to prolong survival with an acceptable QOL
4. Performance status: Lansky or Karnofsky ≥ 50%
5. ORGAN FUNCTION CRITERIA Bone Marrow Function

   * Peripheral ANC ≥ 1.5x109/L; Plt ≥ 100x109/L and Hgb ≥ 80 g/L (RBC transfusion permitted) Renal Function
   * Measured creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73 m2, OR a serum creatinine based on age/gender that meets the criteria outlined in the protocol
   * Urinalysis negative for protein, urine protein:creatinine ratio of ≤ 1, OR a 24-hour urine protein < 1000 mg/dL
   * <Gr.1 abnormalities of K, Ca (confirmed by ionized Ca),Mg or Ph (supplementation allowed) Liver Function
   * Total serum bilirubin ≤ 1.5xULN for age
   * SGPT (ALT) ≤ 2.5 x ULN and SGOT (AST) ≤ 2.5 x ULN
   * Serum albumin ≥ 20 g/L Cardiac Function
   * Adequate systolic ventricular function (LVSF≥ 27% or LVEF ≥ 50%)
   * QTc measured by ECG must be < 450 msec.
   * No history of MI, severe or unstable angina, peripheral vascular disease, or familial QTc prolongation Blood Pressure
   * Blood pressure ≤ 95th percentile for age, height, gender AND one of:
   * No current anti-hypertensive therapy, OR on stable doses of no more than one anti-hypertensive medication CNS Function
   * Subjects with known history of seizures must have well-controlled seizures and not receiving enzyme-inducing anti-convulsants Coagulation Function
   * INR ≤ 1.2 and PTT ≤ 1.2xULN
6. Prior Therapy

   * Myelosuppressive chemo must not have been given within 3 weeks of study enrolment (6 weeks if nitrosourea)
   * At least 7 days must have elapsed since completion of therapy with a growth factor that supports platelet or white cell number or function. At least 14 days must have elapsed after receiving pegfilgrastim.
   * Biologic anti-neoplastic agent (including VEGF-blocking TKI) must not have been administered within 7 days of study enrolment
   * At least 3 half lives of the monoclonal antibody must have elapsed since the last dose administered
   * ≥ 2 weeks must have elapsed since local palliative XRT (small port); > 13 weeks since prior total body irradiation (TBI), craniospinal XRT or > 50% radiation of pelvis; or > 6 weeks if other substantial bone marrow irradiation
   * ≥ 8 weeks must have elapsed since MIBG therapy for neuroblastoma
   * At least 60 days must have elapsed from autologous or allogeneic stem cell transplant with no signs of GVHD.
   * At least 28 days from major surgery and wounds must be healed. At least 7 days from open and/or core biopsy.
7. Ability to take liquid medication by mouth

EXCLUSION:

1. Patients with CNS tumours or known CNS metastases
2. Pregnancy, breast feeding, or unwillingness to use effective contraception during the study
3. Subjects currently receiving:

   * Corticosteroids who haven't been on a stable or decreasing dose of corticosteroid for 7 days prior
   * Another investigational drug; other anti-cancer agents or radiation therapy
   * More than one medication for blood pressure control
   * Therapeutic anticoagulation, including systemic use of warfarin, heparin, or low molecular weight heparin at any dose
   * Aspirin, and/or ibuprofen, or other NSAIDs
   * Drugs metabolized through several of the specific P450 cytochrome isoforms and those receiving drugs with a known risk of torsades de pointes
   * Subjects who require thyroid replacement therapy are not eligible if they have not been receiving a stable replacement dose for at least 4 weeks prior to study enrolment.
4. Subjects who have an uncontrolled infection or serious non-healing would, ulcer or bone fracture.
5. Evidence of active bleeding, intratumoral haemorrhage, or bleeding diathesis, hemoptysis or any evidence of GI hemorrhage.
6. History (within 26 weeks prior to study enrolment) of arterial thromboembolic events (including TIA, CVA, or MI), pulmonary embolism, DVT or other venous thromboembolic event.
7. Evidence of tumour-related or other thrombus at time of enrolment
8. Major surgical procedure, laparoscopic procedure or significant traumatic injury within 28 days prior to Day 1 therapy. Open or core biopsy within 7 days prior to Day 1 of therapy. Fine needle aspirate within 48 hours prior to Day 1 therapy.
9. Previous, documented hypersensitivity reactions to topotecan or pazopanib
10. History of abdominal fistula, GI perforation, or intra-abdominal abscess within 28 days of study enrolment.
11. QTc > 450msec on baseline ECG or history of familial prolonged QTc syndrome
12. History of inflammatory lung disease secondary to exposure to mTOR or tyrosine kinase inhibitors.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of low dose metronomic (LDM)Topotecan | Dose limiting toxicities (DLT) will be identified during the first cycle of therapy (28 days)
  MTD is dependent on the number of subjects who experience a DLT at a given dose level
Recommended phase 2 dose (RP2D) of LDM Topotecan | Dose limiting toxicities (DLT) will be identified during the first cycle of therapy (28 days)
  The RP2D will be defined as the highest dose, at or below the MTD, at which the median number of cycles tolerated by subjects is ≥ 3.

SECONDARY OUTCOMES:
Anti-tumour activity of LDM Topotecan in combination with Pazopanib | 24 months
  To preliminarily define the anti-tumour activity of LDM Topotecan in combination with pazopanib in pediatric solid tumours within the confines of a phase 1 study, and more specifically in cohorts of children with i) neuroblastoma and ii) rhabdomyosarcoma
Pharmacokinetics of LDM Topotecan and Pazopanib | 24 months
  To characterize the pharmacokinetics of LDM Topotecan and Pazopanib, as well as any drug-drug interactions
Anti-angiogenic activity of LDM Topotecan and Pazopanib | 24 months
  To assess the anti-angiogenic activity of this regimen by evaluating changes in plasma cytokines and angiogenic factors (CAF).

CONTACTS AND LOCATIONS:
Overall Officials: Jim Whitlock, Study Chair — The Hospital for Sick Children
Locations (10):
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital, London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - CHU St. Justine Hopital, Montreal, Quebec